CLINICAL TRIAL: NCT06741943
Title: A Prospective, Multicenter, Open-label Study Evaluating an Insulin Pump (model: AR-B200A) for Time in Range (TIR) in Patients with Type 1 Diabetes
Brief Title: Evaluating an Insulin Pump for Time in Range (TIR) in Patients with Type 1 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tao Yuan，MD (Other)
Collaborators: Second Xiangya Hospital of Central South University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor-Investigator, Tao Yuan，MD, Clinical Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR-B200-202401
Record Dates: First submitted 2024-12-07; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes Mellitus; Insulin Pump; Time in Range
Keywords: type 1 diabetes; insulin pump; time in range
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Infusion Systems; Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Insulin pump therapy (Experimental): Subject wearing insulin pump (model: AR-B200A) and continuous glucose monitoring (FreeStyle Libre)
  Interventions: Device: insulin pump (model: AR-B200A)

INTERVENTIONS:
Device: insulin pump (model: AR-B200A) — USE insulin pump (model: AR-B200A) and continuous glucose monitoring (FreeStyle Libre)
  Other Names: AR-B200A; FreeStyle Libre; insulin pump; continuous glucose monitoring

SUMMARY:
Diabetes mellitus is a metabolic disorder caused by genetic, environmental changes, mental health issues, immune disorders, and other factors. It may occur with or without insulin resistance, insulin secretion defect, or impaired biological function of insulin. The condition is characterized by chronic hyperglycemia and targeted damage to multiple systems and organs. Insulin pump therapy is an advanced method for managing diabetes that mimics the natural secretion of insulin by providing continuous delivery to diabetic patients. Compared to traditional multiple injections, the use of an insulin pump reduces the number of injections required and improves patient compliance and treatment convenience. The medical team can customize the insulin pump treatment based on each patient's specific situation in order to achieve optimal blood sugar control and effectively reduce the risk of complications. In recent years, there has been significant attention given to glucose-in-target time (TIR), which refers to the amount of time blood sugar levels are within a range of 3.9 to 10.0 mmol/L in non-pregnant adults measured either as minutes or as a percentage (%). This clinical trial aims to collect data on using an insulin pump (Model: AR-B200A) combined with a scanning glucose monitoring system (Model: FreeStyle Libre, 20163072472) for continuous subcutaneous insulin infusion in type 1 diabetes patients in order to provide reference for related clinical applications.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled:

1. Age between 8 and 75 years old, regardless of gender;
2. Subjects with T1DM (including adult occult autoimmune diabetes mellitus (LADA)) who have been judged by investigators to require insulin pump therapy;
3. Subjects who are able to cooperate with insulin pump therapy and derive weekly data from insulin pump during study treatment;
4. During the study period, the subject's total daily insulin should be ≥8 units;
5. Subjects who are able to follow a diabetic diet;
6. Those who can voluntarily sign informed consent.

Exclusion Criteria:

Subjects are excluded if they meet any of the following criteria:

1. Hyperglycemia with severe circulatory disorders and shock;
2. Acute complications of diabetes (such as diabetic ketoacidosis, diabetic hyperosmolar non-ketotic coma);
3. A history of 2 or more episodes of severe hypoglycemia leading to medical assistance, coma or seizure in the 6 months prior to screening;
4. The presence of at least 4 hypoglycemic symptoms, occurrence or detection of hypoglycemic events within 1 month before screening;
5. Patients with hyperthyroidism;
6. Any serious systemic disease determined by the investigator or any other disease that the investigator believes may interfere with the results of this study, including but not limited to mental illness, immune system disease, malignancy, etc.;
7. Patients who developed the following cardiac conditions in the 6 months prior to screening: a) decompensated cardiac insufficiency (New York College of Cardiology (NYHA) Class III or IV); b) unstable angina; c) History of myocardial infarction, coronary artery bypass grafting, or coronary stent implantation; d) Uncontrolled or severe arrhythmia;
8. Patients with the following cerebrovascular diseases in the 6 months before screening: a) transient ischemic attack; b) stroke;
9. Subjects with sickle cell anaemia, thalassaemia or hemoglobinopathy;
10. Subjects who have received, or plan to receive, red blood cell transfusions or erythropoietin (EPO) therapy within the 3 months prior to screening;
11. Used immunosuppressants, cytotoxic drugs, systemic steroid drugs (excluding topical or inhaled preparations) for more than 7 days in the 3 months prior to screening or planned to be used during the study period;
12. Screening subjects who have used hormone therapy for 3 or more consecutive days in the preceding 3 months, are currently using, or plan to use systemic hormone therapy during the study period;
13. Present with known proliferative retinal lesions or other history of visual impairment;
14. History of hearing loss;
15. Impaired liver and kidney function (total bilirubin > 1.5 times the upper limit of normal, alanine aminotransferase (ALT) > 2.5 times the upper limit of normal; Glomerular filtration rate (eGFR) < 30 mL/min/1.73m2);
16. Subjects with erythrocyte specific volume lower than the lower limit of normal laboratory values;
17. Patients with abnormal coagulation function (activated partial thromboplastin time (APTT) or prothrombin time (PT) test results >1.5 times the upper limit of normal value);
18. Participants who plan to use drugs containing acetaminophen, vitamin C, etc. that affect blood glucose measurement during the study period;
19. Major surgery is planned during the study period and will directly affect subjects treated with insulin pumps;
20. Subjects who do not have self-glucose monitoring conditions or do not accept home self-glucose monitoring;
21. People who are allergic to glucose sensors, subcutaneous infusion sets, and medical tape;
22. There are adverse skin conditions (such as diffuse subcutaneous nodules, psoriasis, rash, staphylococcal infection, psoriasis, scars, stretch marks, etc.) at the site where the glucose sensor and insulin pump subcutaneous infusion device are planned to be placed;
23. Subjects who are unwilling to bury the infusion tube subcutaneously or wear the pump for a long time, and psychologically do not accept insulin pump treatment;
24. Subjects and their families lacked relevant knowledge and were unable to correctly master the user after receiving training (excluding subjects who were hospitalized or admitted to the hospital during the study period for insulin pump operation by a doctor/nurse);
25. Subjects with poor compliance, unable to cooperate with intensive treatment or irregular exercise;
26. Young or elderly subjects who are unable to take care of themselves and have no guardian;
27. Subjects who are not able to use effective contraception during pregnancy, lactation or during the study;
28. Participated in other clinical trials within 3 months prior to screening;
29. Other conditions deemed unsuitable for inclusion by the researcher.

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time in range (TIR) at week 4 of treatment | week 4 ±3 days of treatment
  TIR is defined as the percentage (%) of the entire day that is within the target range of blood sugar (3.9 to 10.0 mmol/L) [1], measured in minutes.
  The mean of CGM monitoring for 3 days prior to participation in the V9 visit (week 4 ±3 days of treatment) (excluding the day of follow-up) was used as TIR at week 4 of treatment. The basic principle is to choose 3 days close to the date of the visit. If blood glucose monitoring was not possible for 1 of the 3 days close to the visit date, the data of the previous 1 day was used instead; If blood glucose monitoring was not possible for 2 out of 3 days close to the visit date, data from 2 days ahead was used instead.

SECONDARY OUTCOMES:
Hemoglobin a1c (HbA1c) | from baseline at week 4 and week 1 after treatment
  HbA1c (%, mmol/mol) and its change from baseline at week 4 and week 1 after treatment were recorded.
Glycated albumin (GA) | from baseline at week 1, week 2, week 4 and week 1 after treatment
  GA (%, g/dL) and its change from baseline at week 1, week 2, week 4 and week 1 after treatment were recorded.
Time in Range (TIR), time below range (TBR), time above range (TAR) | through study completion, an average of 3 month
  TBR: Time below the blood glucose target range (3.9 to 10.0 mmol/L). TAR: Time above the target blood glucose range (3.9 to 10.0 mmol/L).
TIR, TBR and TAR all reached the control target | at week 1, week 2, week 4 and week 1 after treatment
  The proportion of subjects whose TIR, TBR and TAR all reached the control goal at week 1, week 2, week 4 and week 1 after treatment was calculated.
glucose management indicator (GMI) | through study completion, an average of 3 month
  GMI（mmol/mol）=12.71+4.70587×mean glucose
self monitoring of blood glucose (SMBG) blood glucose compliance rate | through study completion, an average of 3 month
  Blood glucose compliance rate means that both fasting blood glucose and postprandial blood glucose are controlled within the target range.
  Control objectives of T1DM subjects: empty abdominal blood glucose 4.0~7.0 mmol/L, postprandial blood glucose 5.0~10.0 mmol/L; The fasting blood glucose was recorded before breakfast and the postprandial blood glucose was recorded 2 hours after three meals.
Blood lipid | changes from baseline were recorded at week 1, week 2, week 4 and week 1 after treatment
  The blood lipid levels (triglyceride (TG), total cholesterol (TC), high density lipoprotein (HDL-C), low density lipoprotein (LDL-C)) and their changes from baseline were recorded at week 1, week 2, week 4 and week 1 after treatment
weight(kg) | baseline period, the first week of treatment, the second week, the fourth week, the first week after treatment
  The baseline period (kg), the first week of treatment (kg) , the second week (kg), the fourth week (kg), the first week after treatment and the change from baseline were recorded.
Insulin pump infusion volume | through study completion, an average of 3 month
  Total Daily Base Rate Infusion = Total Daily Infusion - Total daily high dose
Instrument performance evaluation | through study completion, an average of 3 month
  On the first day and the fourth week of treatment, the actual operator (doctor/nurse/subject/subject's family) completed the performance evaluation of the device, including "identification", "operation", "product stability" and "overall design", and the score of each item was 0 to 10 points, 0 points indicated dissatisfaction and 10 points indicated very satisfaction.
Diabetes Treatment Satisfaction Questionnaire-status(DTSQS) | at baseline, week 4 of treatment
  Participants completed the Diabetes Treatment Satisfaction Questionnaire-status(DTSQS)at baseline, week 4 of treatment（the higher scores mean a better outcome.）
Insulin Pump Satisfaction Questionnaire | at baseline, week 4 of treatment
  Participants completed insulin pump satisfaction questionnaires at day 1 and week 4 of treatment（the higher scores mean a better outcome.）
Exercise | through study completion, an average of 3 month
  After signing the informed consent form, the subjects began to record their daily exercise type and duration (in minutes(min)).
  If the subjects did exercise, they were required to record the exercise situation in time, including the exercise date, weight, exercise start time, exercise treatment method (walking, running, cycling, swimming, etc.) and exercise duration (in minutes(min)).
mean glucose（MG） | through study completion, an average of 3 month
  Average daily blood glucose of subjects (mmol/l)
standard deviation (SD) | through study completion, an average of 3 month
  Standard deviation of daily blood glucose in subjects (mmol/l)
coefficient of variation (CV) | through study completion, an average of 3 month
  Daily blood glucose coefficient of variation (%)
Mean Amplitude of Glucose Exposure (MAGE) | through study completion, an average of 3 month
  Daily blood glucose mean amplitude of glucose exposure (mmol/l)
BMI （kg/m^2） | baseline period, the first week of treatment, the second week, the fourth week, the first week after treatment
  The baseline period , the first week of treatment , the second week , the fourth week , the first week after treatment and the change from baseline were recorded.
Diet | through study completion, an average of 3 month
  After signing the informed consent form, the subjects began to record their daily diet(Carbohydrates and other foods,in grams(g)) .
  Records of daily meals include: date of meals, number of meals (breakfast, lunch, dinner, and extra meals), time of meal (from the first bite), and type of meals eaten (staples, vegetables, fruits, meat, eggs, dairy, nuts, desserts, and others). Note: Before eating, the subjects took photos of the food (vertically overhead) and provided the photos to the research center.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No